CLINICAL TRIAL: NCT02334800
Title: A Phase 1, Open-label, Single Dose, Parallel-cohort Study To Evaluate The Pharmacokinetics Of Palbociclib (Pd-0332991) In Subjects With Impaired Hepatic Function
Brief Title: A Study To Describe The Effect Of Impaired Hepatic Function Of The Pharmacokinetics Of Palbociclib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A5481013
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2017-05

CONDITIONS: Healthy, Hepatic Insufficiency
Keywords: Palbociclib, PD-0332991, Hepatic Impairment
MeSH Terms: conditions — Hepatic Insufficiency | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Volunteers (Experimental): Cohort of Healthy Volunteers
  Interventions: Drug: Palbociclib 75 mg Capsule
- Mild Hepatic Impairment (Experimental): Cohort of mild hepatic impairment subjects meeting the criteria for Child-Pugh Class A
  Interventions: Drug: Palbociclib 75 mg Capsule
- Moderate Hepatic Impairment (Experimental): Cohort of moderate hepatic impairment subjects meeting the criteria for Child-Pugh Class B
  Interventions: Drug: Palbociclib 75 mg Capsule
- Severe Hepatic Impairment (Experimental): Cohort of severe hepatic impairment subjects meeting the criteria for Child-Pugh Class C
  Interventions: Drug: Palbociclib 75 mg Capsule

INTERVENTIONS:
Drug: Palbociclib 75 mg Capsule — Single oral 75 mg dose of palbociclib followed by serial PK sampling up to 192 hours post-dose (up to 120 hours post-dose for the healthy volunteer cohort).
  Other Names: Palbociclib, PD-0332991

SUMMARY:
This is a phase 1 study to describe the plasma pharmacokinetics of a single oral 75mg dose of palbociclib administered to healthy volunteers, and subjects with mild, moderate, and severely impaired hepatic function.

DETAILED DESCRIPTION:
This is a 4-cohort single period study. The four cohorts will consist of healthy volunteers, and subjects with mild, moderate, and severely impaired hepatic function. Each cohort will receive the same treatment consisting of a single oral 75mg dose of palbociclib administered with food. Serial PK samples will be drawn up to 120 hours post dose for the cohort consisting of healthy volunteers, and will continue until up to 192 hours post-dose for the cohorts of hepatic impairment subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18 to 40 kg/m2; and a total body weight >50 kg (110 lbs)
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy)
* A positive urine drug screen
* Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential; male subjects with partners currently pregnant; male subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception for the duration of the study and for 90 days after the last dose of investigational product
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Blood donation of approximately 1 pint (500 mL) or more within 56 days prior to dosing
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol
* Use of tobacco or nicotine products in excess of 5 cigarettes per day (or equivalent)
* History of sensitivity to palbociclib

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2016-10-09 (Actual); Study Completion 2016-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Weston Diagnostics (Ultrasound Facility), Orlando, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481013&StudyName=A%20Phase%201%2C%20Open-label%2C%20Single%20Dose%2C%20Parallel-cohort%20Study%20To%20Evaluate%20The%20Pharmacokinetics%20Of%20Palbociclib%20%28pd-0332991%29%20In%20Subjects%20With%20Impaired%20Hepatic%20Function

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 28 participants were assigned to and received the study treatment (7 participants in each cohort).
Groups:
- Palbociclib 75 mg (Normal Hepatic Function, Cohort 1): Participants with normal hepatic function were enrolled in this cohort. Participants received single oral dose of palbociclib 75 mg approximately 10 minutes after completion of the moderate fat standard calorie breakfast, with approximately 240 mL of ambient temperature water.
- Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2): Participants with Child-Pugh scores of 5 to 6 points were enrolled in this cohort. Participants received single oral dose of palbociclib 75 mg approximately 10 minutes after completion of the moderate fat standard calorie breakfast, with approximately 240 mL of ambient temperature water.
- Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3): Participants with Child-Pugh scores of 7 to 9 points were enrolled in this cohort. Participants received single oral dose of palbociclib 75 mg approximately 10 minutes after completion of the moderate fat standard calorie breakfast, with approximately 240 mL of ambient temperature water.
- Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4): Participants with Child-Pugh scores of 10 to 15 points were enrolled in this cohort. Participants received single oral dose of palbociclib 75 mg approximately 10 minutes after completion of the moderate fat standard calorie breakfast, with approximately 240 mL of ambient temperature water.
Period: Overall Study
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Started | 7 | 7 | 7 | 7
Received Treatment | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4) | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (2.6) | 53.9 (5.1) | 57.9 (4.2) | 57 (5.3) | 56.6 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 4 | 10
  Male | 4 | 6 | 5 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinite Time (AUCinf)
Description: AUCinf is area under the plasma concentration time curve from time 0 extrapolated infinite time. It is calculated as AUClast + (Clast/kel), where AUClast is area under the concentration-time curve from time 0 to the time of the last quantifiable concentration, Clast is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose for all participants. Additional pharmacokinetics samples were collected from participants in hepatic impairment cohorts (Cohorts 2, 3 and 4) at 144, 168, and 192 hours post-dose.
Population: The pharmacokinetics parameter analysis population was defined as all participants enrolled and treated who had at least 1 of the palbociclib pharmacokinetics parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
nanogram*hour/milliliter (ng*hr/mL) | 1031 (24) | 758.9 (31) | 1189 (22) | 1378 (29)
Statistical Analysis 1: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2); Test type: Superiority or Other; ratio of adjusted geometric mean = 73.60, 90% CI 2-sided [57.81 to 93.71]
Statistical Analysis 2: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3); Test type: Superiority or Other; ratio of adjusted geometric mean = 115.30, 90% CI 2-sided [90.57 to 146.79]
Statistical Analysis 3: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4); Test type: Superiority or Other; ratio of adjusted geometric mean = 133.68, 90% CI 2-sided [105.00 to 170.19]

2. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Cmax is maximum plasma concentration. It is observed directly from data.
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose for for all participants. Additional pharmacokinetics samples were collected from participants in hepatic impairment cohorts (Cohorts 2, 3 and 4) at 144, 168, and 192 hours post-dose.
Population: The pharmacokinetics concentration population was defined as all participants enrolled and treated who had at least 1 palbociclib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
nanogram/milliliter (ng/mL) | 28.64 (20) | 27.20 (37) | 33.72 (28) | 37.20 (48)
Statistical Analysis 1: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2); Test type: Superiority or Other; ratio of adjusted geometric mean = 94.99, 90% CI 2-sided [69.93 to 129.03]
Statistical Analysis 2: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3); Test type: Superiority or Other; ratio of adjusted geometric mean = 117.75, 90% CI 2-sided [86.69 to 159.95]
Statistical Analysis 3: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4); Test type: Superiority or Other; ratio of adjusted geometric mean = 129.89, 90% CI 2-sided [95.63 to 176.43]

3. Secondary Outcome: Unbound AUCinf (AUCinf,u)
Description: AUCinf,u is unbound AUCinf, where AUCinf is area under the concentration-time curve from time 0 extrapolated to infinite time. It is obtained by fu*AUCinf, where fu is the fraction of unbound drug in plasma.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng*hr/mL | 196.6 (26) | 163.2 (32) | 264.1 (25) | 347.8 (23)
Statistical Analysis 1: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2); Test type: Superiority or Other; ratio of adjusted geometric mean = 83.01, 90% CI 2-sided [65.37 to 105.43]
Statistical Analysis 2: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3); Test type: Superiority or Other; ratio of adjusted geometric mean = 134.28, 90% CI 2-sided [105.73 to 170.53]
Statistical Analysis 3: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4); Test type: Superiority or Other; ratio of adjusted geometric mean = 176.88, 90% CI 2-sided [139.28 to 224.63]

4. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast)
Description: AUClast is area under the plasma concentration time curve from time 0 to time of last quantifiable concentration. It is obtained from linear/log trapezoidal method.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng*hr/mL | 973.3 (24) | 708.6 (34) | 1125 (24) | 1311 (31)
Statistical Analysis 1: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2); Test type: Superiority or Other; ratio of adjusted geometric mean = 72.81, 90% CI 2-sided [56.43 to 93.93]
Statistical Analysis 2: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3); Test type: Superiority or Other; ratio of adjusted geometric mean = 115.57, 90% CI 2-sided [89.58 to 149.11]
Statistical Analysis 3: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4); Test type: Superiority or Other; ratio of adjusted geometric mean = 134.66, 90% CI 2-sided [104.38 to 173.73]

5. Secondary Outcome: Unbound AUClast (AUClast,u)
Description: AUClast,u is unbound AUClast, where AUClast is area under the concentration-time curve from time 0 to the time of the last quantifiable concentration. It is obtained by fu*AUClast, where fu is the fraction of unbound drug in plasma.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng*hr/mL | 185.5 (26) | 152.4 (35) | 250.3 (26) | 331.0 (24)
Statistical Analysis 1: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2); Test type: Superiority or Other; ratio of adjusted geometric mean = 82.14, 90% CI 2-sided [63.83 to 105.71]
Statistical Analysis 2: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3); Test type: Superiority or Other; ratio of adjusted geometric mean = 134.90, 90% CI 2-sided [104.82 to 173.60]
Statistical Analysis 3: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4); Test type: Superiority or Other; ratio of adjusted geometric mean = 178.39, 90% CI 2-sided [138.62 to 229.57]

6. Secondary Outcome: Apparent Clearance After Oral Dose(CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance is obtained by dose/AUCinf, where AUCinf is the area under the concentration-time curve from time 0 extrapolated to infinite time.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour (L/hr)
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
liter/hour (L/hr) | 72.64 (24) | 98.84 (31) | 63.15 (22) | 54.42 (29)

7. Secondary Outcome: Unbound CL/F (CLu/F)
Description: CLu/F is unbound CL/F, where CL/F is apparent clearance after oral dose. It is obtained by dose/AUCinf,u, where AUCinf,u is unbound AUCinf (area under the concentration-time curve from time 0 extrapolated to infinite time).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
L/hr | 381.3 (26) | 459.2 (32) | 283.8 (25) | 215.8 (23)

8. Secondary Outcome: Unbound Cmax (Cmax,u)
Description: Cmax,u is unbound Cmax, where Cmax is maximum plasma concentration. It is obtained by fu*Cmax, where fu is fraction of unbound drug in plasma.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL | 5.456 (23) | 5.858 (37) | 7.501 (34) | 9.399 (47)
Statistical Analysis 1: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2); Test type: Superiority or Other; ratio of adjusted geometric mean = 107.37, 90% CI 2-sided [78.06 to 147.68]
Statistical Analysis 2: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3); Test type: Superiority or Other; ratio of adjusted geometric mean = 137.50, 90% CI 2-sided [99.96 to 189.12]
Statistical Analysis 3: Comparison: Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) vs Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4); Test type: Superiority or Other; ratio of adjusted geometric mean = 172.27, 90% CI 2-sided [125.25 to 236.96]

9. Secondary Outcome: Fraction of Unbound Drug in Plasma (fu)
Description: Fu is the fraction of unbound drug in plasma. It is obtained from measurement of protein binding.
Time Frame: Eight (8) hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
ratio | 0.1910 (0.015) | 0.2157 (0.014) | 0.2236 (0.025) | 0.2546 (0.036)

10. Secondary Outcome: Terminal Half-Life (t1/2)
Description: T1/2 is terminal half-life. It is obtained by loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour (hr)
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
hour (hr) | 25.84 (4.22) | 27.23 (5.49) | 35.03 (4.61) | 33.84 (5.39)

11. Secondary Outcome: Time for Cmax (Tmax)
Description: Tmax is time for maximum plasma concentration. It is observed directly from data as time of first occurrence of maximum plasma concentration.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
hr | 8.00 [6.00 to 12.0] | 6.00 [6.00 to 6.00] | 6.00 [2.00 to 6.00] | 6.00 [2.00 to 8.00]

12. Secondary Outcome: Apparent Volunm of Distribution After Oral Dose (Vz/F)
Description: Vz/F is the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. It is influenced by the fraction absorbed. It is obtained by dose/(AUCinf•kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve, and AUCinf is the area under the concentration-time curve from time 0 extrapolated to infinite time.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
liter (L) | 2679 (18) | 3814 (36) | 3168 (26) | 2627 (29)

13. Secondary Outcome: Unbound Vz/F (Vz,u/F)
Description: Vz,u/F is unbound Vz/F, where Vz/F is apparent volume of distribution after oral dose. It is obtained by dose/(AUCinf,u*kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve, and AUCinf,u is unbound AUCinf (area under the concentration-time curve from time 0 extrapolated to infinite time).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
L | 14060 (24) | 17730 (36) | 14260 (32) | 10410 (30)

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Any events occurring following start of treatment or increasing in severity are counted as treatment emergent. Relatedness to palbociclib is assessed by the investigator (Yes/No). Participants with multiple occurrences of an adverse event within a category are counted once within the category.
Time Frame: Adverse events were recorded on the Case Report Form from the time the participant had taken at least 1 dose of palbociclib through the participant's last visit.
Population: All participants who received at least 1 dose of study medication were included in the safety analyses and listings.
Measure: Number; unit: participant
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
participant | 2 | 0 | 2 | 1

15. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events
Description: A serious adverse event is any untoward medical occurrence at any dose that resulted in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; or results in congenital anomaly/birth defect. Any events occurring following start of treatment or increasing in severity are counted as treatment emergent. Relatedness to palbociclib is assessed by the investigator (Yes/No).
Time Frame: The active reporting period for serious adverse events began from the time that the participant provided informed consent through and including 28 calendar days after the last administration of palbociclib.
Population: All participants who received at least 1 dose of study medication were included in the safety analyses and listings.
Measure: Number; unit: participant
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
participant | 0 | 0 | 1 | 0

16. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory tests included tests that were performed under the categories of hematology, chemistry, urinalysis, other, and additional tests needed for Hy's law.
Time Frame: Baseline up to Day 6 for Cohort 1 and to Day 9 for Cohorts 2, 3, and 4, inclusive of baseline values.
Population: All participants who received at least 1 dose of study medication were included in the safety analyses and listings.
Measure: Number; unit: participants
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
participants | 6 | 6 | 5 | 7

17. Secondary Outcome: Number of Participants With Physical Examination Test Abnormalities (Change From Prior Visit)
Description: A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The limited or abbreviated physical examination was focused on general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms.
Time Frame: Baseline up to Day 6 for Cohort 1 and to Day 9 for Cohorts 2, 3, and 4.
Population: All participants who received at least 1 dose of study medication were included in the safety analyses and listings.
Measure: Number; unit: participant
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
participant | 0 | 0 | 2 | 0

18. Secondary Outcome: Number of Participants With Post Baseline Vital Signs Values Meeting Categorical Summarization Criteria
Description: The number of participants with post baseline vital signs values meeting the following criteria was reported: A. absolute value of supine systolic blood pressure less than (<) 90 mmHg; B. absolute value of diastolic blood pressure <50 mmHg; C. absolute value of supine pulse rate <40 bmp; D. absolute value of supine pulse rate larger than (>) 120 bmp; E. maximum increase from baseline in supine systolic blood pressure larger than and equal to (>=) 30 mmHg; F. maximum increase from baseline in supine diastolic blood pressure >=20 mmHg; G. maximum decrease from baseline in supine systolic blood pressure >=30 mmHg; and H. maximum decrease from baseline in supine diastolic blood pressure >=20 mmHg.
Time Frame: Baseline up to Day 6 for Cohort 1 and to Day 9 for Cohorts 2, 3, and 4, not including baseline values.
Population: All participants who received at least 1 dose of study medication were included in the safety analyses and listings.
Measure: Number; unit: participant
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
participant
  criterion A | 0 | 1 | 0 | 0
  criterion B | 0 | 0 | 0 | 2
  criterion C | 0 | 0 | 0 | 0
  criterion D | 0 | 0 | 0 | 0
  criterion E | 0 | 0 | 0 | 0
  criterion F | 0 | 0 | 0 | 0
  criterion G | 0 | 0 | 1 | 1
  criterion H | 0 | 0 | 0 | 1

19. Secondary Outcome: Number of Participants With Post Baseline Electrocardiogram Values Meeting Categorical Summarization Criteria (Maximum Absolute Values)
Description: Maximum absolute values of post baseline electrocardiogram were summarized for PR interval, QRS complex, QT interval, QTcB (QT interval calculated using Bazett's correction factor), and QTcF (QT interval calculated using Fridericia's correction factor). The number of participants with maximum absolute values of post baseline electrocardiogram meeting the following criteria was reported: (1) PR interval >=300 msec; (2) QRS complex >=140 msec; (3) QT interval 450 to <480 msec; (4) QT interval 480 to <500 msec; (5) QT interval >= 500 msec; (6) QTcB 450 to <480 msec; (7) QTcB 480 to <500 msec; (8) QTcB >= 500 msec; (9) QTcF 450 to <480 msec; (10) QTcF 480 to <500 msec; and (11) QTcF >=500 msec. Seven (7) participants in each cohort were evaluated for electrocardiogram tests except that 6 participants in the moderate hepatic impairment cohort (Cohort 3) were evaluated for PR interval.
Time Frame: Baseline up to Day 6 for Cohort 1 and to Day 9 for Cohorts 2, 3, and 4, not including baseline values.
Population: All participants who received at least 1 dose of study medication were included in the safety analyses and listings. Seven (7) participants in each cohort were evaluated for electrocardiogram tests except that 6 participants in the moderate hepatic impairment cohort (Cohort 3) were evaluated for PR interval.
Measure: Number; unit: participant
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
participant
  PR interval >=300 msec | 0 | 0 | 0 | 0
  QRS complex >=140 msec | 0 | 0 | 0 | 0
  QT interval 450 to <480 msec | 0 | 1 | 1 | 4
  QT interval 480 to <500 msec | 0 | 2 | 0 | 0
  QT interval >= 500 msec | 0 | 0 | 0 | 0
  QTcB 450 to <480 msec | 0 | 1 | 2 | 2
  QTcB 480 to <500 msec | 0 | 0 | 0 | 3
  QTcB >= 500 msec | 0 | 0 | 0 | 0
  QTcF 450 to <480 msec | 0 | 1 | 0 | 5
  QTcF 480 to <500 msec | 0 | 0 | 0 | 0
  QTcF >=500 msec | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Post Baseline Electrocardiogram Values Meeting Categorical Summarization Criteria (Maximum Increase From Baseline)
Description: Maximum increases from baseline for post baseline electrocardiogram values were summarized for PR interval, QRS complex, QT interval, QTcB (QT interval calculated using Bazett's correction factor), and QTcF (QT interval calculated using Fridericia's correction factor). The number of participants with maximum increase from baseline for post baseline electrocardiogram values meeting the following criteria was reported: (1) percent change of PR interval >=25/50%; (2) percent change of QRS complex >=50%; (3) QT interval 30 to <60 msec; (4) QT interval >= 60 msec; (5) QTcB 30 to <60 msec; (6) QTcB >= 60 msec; (7) QTcF 30 to <60 msec; and (8) QTcF >= 60 msec. Seven (7) participants in each cohort were evaluated for electrocardiogram tests except that 6 participants in the moderate hepatic impairment cohort (Cohort 3) were evaluated for PR interval.
Time Frame: Baseline up to Day 6 for Cohort 1 and to Day 9 for Cohorts 2, 3, and 4, not including baseline values.
Population: as for outcome 19
Measure: Number; unit: paticipant
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
paticipant
  percent change of PR interval >=25/50% | 0 | 0 | 0 | 0
  percent change of QRS complex >=50% | 0 | 0 | 0 | 0
  QT interval 30 to <60 msec | 0 | 0 | 0 | 2
  QT interval >= 60 msec | 0 | 0 | 0 | 0
  QTcB 30 to <60 msec | 0 | 0 | 0 | 1
  QTcB >= 60 msec | 0 | 0 | 0 | 1
  QTcF 30 to <60 msec | 0 | 0 | 0 | 0
  QTcF >= 60 msec | 0 | 0 | 0 | 1

21. Secondary Outcome: Number of Participants With Concomitant Medications
Description: Treatments taken after the first dose of study treatment were documented as concomitant treatments.
Time Frame: From screening through and including Day 6 for Cohort 1, and from screening through and including Day 9 for Cohorts 2, 3, and 4.
Population: All participants who received at least 1 dose of study medication were included in the safety analyses and listings.
Measure: Number; unit: participant
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Number analyzed (Participants) | 7 | 7 | 7 | 7
participant | 0 | 3 | 7 | 7

ADVERSE EVENTS:
Time Frame: For adverse event, from the time participant took at least 1 dose of palbociclib through the last visit. For serious adverse event, from the participant provided informed consent through 28 calendar days post last administration of palbociclib.
Description: The listing of Other Adverse Events does not include events already captured in the Serious Adverse Event listing. An adverse event of diarrhea was reported in the moderate hepatic impairment cohort after database lock and release. It was therefore not recorded in the clinical database, but was added here for completeness and transparency.
Arm/Group | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 1/7 | 0/7
Other Adverse Events (participants affected / at risk) | 2/7 | 0/7 | 2/7 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) (N=7) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) (N=7) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) (N=7) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4) (N=7)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib 75 mg (Normal Hepatic Function, Cohort 1) (N=7) | Palbociclib 75 mg (Mild Hepatic Impairment, Cohort 2) (N=7) | Palbociclib 75 mg (Moderate Hepatic Impairment, Cohort 3) (N=7) | Palbociclib 75 mg (Severe Hepatic Impairment, Cohort 4) (N=7)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Infusion site bruising (General disorders) | 0 | 0 | 1 | 0
Infusion site reaction (General disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Radial nerve compression (Nervous system disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.